CLINICAL TRIAL: NCT01690364
Title: Comparison of the Effects of Vecuronium and Cisatracurium on Electrophysiologic Monitoring During Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Jin Lee, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2012-05-090-001
Record Dates: First submitted 2012-09-10; First posted 2012-09-21 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Motor Evoked Potential Monitoring; General Anesthesia; Neurosurgery; Brain Tumor; Spine Tumor; Cerebral Aneurysm
Keywords: Motor evoked potential monitoring; General Anesthesia; Neurosurgery; Cisatracurium; Vecuronium
MeSH Terms: conditions — Brain Neoplasms; Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cisatracurium Group (Experimental): MEP monitoring with continuous infusion of cisatracurium during general anesthesia
  Interventions: Other: MEP monitoring with continuous infusion of cisatracurium during general anesthesia
- Vecuronium Group (Active Comparator): MEP monitoring with continuous infusion of vecuronium during general anesthesia
  Interventions: Other: MEP monitoring with continuous infusion of vecuronium during general anesthesia

INTERVENTIONS:
Other: MEP monitoring with continuous infusion of vecuronium during general anesthesia — MEP monitoring with continuous infusion of vecuronium during general anesthesia
  Arms: Vecuronium Group
Other: MEP monitoring with continuous infusion of cisatracurium during general anesthesia — MEP monitoring with continuous infusion of cisatracurium during general anesthesia
  Arms: Cisatracurium Group

SUMMARY:
Recently intraoperative motor evoked potential monitoring (MEP) is widely used to reduce neural damage during neurosurgery.

As neuromuscular blockade(NMB) during MEP monitoring decreases the amplitude of MEP, partial NMB is usually maintained during general anesthesia. Continuous infusion of NMB agent is preferred than bolus infusion during MEP monitoring. There are a lot of NMB agents in clinical use. But there have been no reports about the effect of changing NMB agent on efficacy of MEP monitoring.

Therefore, the investigators performed a randomized controlled trial to evaluate the effect of changing NMB agent on the variability of MEP amplitude during neurosurgery.

DETAILED DESCRIPTION:
Recently intraoperative motor evoked potential monitoring (MEP) is widely used to reduce neural damage during neurosurgery.

As neuromuscular blockade(NMB) during MEP monitoring decreases the amplitude of MEP, partial NMB is usually maintained during general anesthesia. Continuous infusion of NMB agent is preferred than bolus infusion during MEP monitoring. There are a lot of NMB agents in clinical use. But there have been no reports about the effect of changing NMB agent on efficacy of MEP monitoring.

Therefore, the investigators performed a randomized controlled trial to evaluate the effect of changing NMB agent on the variability of MEP amplitude during neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing neurosurgery with intraoperative motor evoked potential monitoring

Exclusion Criteria:

* Patients who can not undergo motor evoked potential monitoring due to central or peripheral neuromuscular disease (e.g. Cerebral palsy, Myasthenia gravis, Acute spinal injury, neurologic shock)
* Patients with hepatic or renal disease with altered metabolism of vecuronium
* Patients with medication which influence the metabolism of vecuronium (e.g. calcium channel blocker, aminoglycoside antibiotics, Lithium, MgSO4)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
MEP amplitude | 15 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 30 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 45 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 60 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 75 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 90 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 105 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 120 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 135 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 150 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 165 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 180 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 195 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 210 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 225 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 240 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 255 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 270 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 285 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude
MEP amplitude | 300 min after anesthetic induction
  intraoperative motor evoked potential monitoring amplitude

SECONDARY OUTCOMES:
Coefficient of variation (CV) of MEP amplitude | at the end of the surgery (5H after the start of surgery)
  Coefficient of variation (CV) of intraoperative motor evoked potential monitoring amplitude
Average of MEP amplitudes | at the end of the surgery (5H after the start of surgery)
  Average of all measured MEP amplitudes in a subject
The frequency of adjusting the infusion dose of muscle relaxant | at the end of the surgery (5H after the start of surgery)
  The frequency of adjusting the infusion dose of muscle relaxant
Average of Latency of MEP amplitude | at the end of the surgery (5H after the start of surgery)
  Average of Latency of MEP amplitude

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea